CLINICAL TRIAL: NCT00229632
Title: A Six Month Double-Blind, Placebo-Controlled Phase 2 Clinical Trial to Determine the Safety and Efficacy of Idebenone Administered to Patients With Friedreich's Ataxia
Brief Title: Idebenone to Treat Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 050245; 05-N-0245
Record Dates: First submitted 2005-09-29; First posted 2005-09-29 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03-14

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich's Ataxia; Idebenone; Ataxia; Drug Trial; Randomized Trial; Friedreich Ataxia; FA
MeSH Terms: conditions — Friedreich Ataxia; Ataxia | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Idebenone — Idebenone is a short-chain benzoquinone derivative of similar structure to ubiquinone (coenzyme Q10). This compound was synthesized and developed initially by Takeda Chemical Industries, Ltd. (Osaka, Japan) and designated as CV-2619. The chemical name for idebenone is 6-(10-Hydroxydecyl)-2,3-dimethoxy-5-methyl-1,4-benxoquinone. Santhera Pharmaceuticals (Liestal, Switzerland) LLC, will supply drug for this study as specified by a clinical trial agreement.

SUMMARY:
This study will determine whether a drug called idebenone is safe and effective in reducing the level of oxidants that are believed to damage the nervous system and hearts in patients with Friedreich's ataxia. Friedreich's ataxia is caused by an abnormality in the gene that makes a protein called frataxin, which is necessary for the proper functioning of energy-producing parts of cells called mitrochondria. In Friedreich's ataxia, the mitochondria become overloaded with iron, and high levels of harmful compounds called oxidants are formed. These oxidants are believed to damage the cells of the nervous system and hearts of people with Friedreich's ataxia. Idebenone is a man-made drug similar to a naturally occurring compound known as Coenzyme Q10. This study will test whether idebenone can alleviate some of the symptoms of Friedreich's ataxia and slow or halt the progression of the disease.

Patients with genetically confirmed Friedreich's ataxia who are between 9 and 18 years of age, weigh between 65 and 175 pounds and can walk 25 feet with or without an assistive device may be eligible for this study. Candidates are screened with blood tests and a review of their medical records.

Participants undergo the following tests and procedures:

* Medical interview and physical examination. Tests include blood and urine tests, an electrocardiogram, or EKG (recording of the electrical activity of the heart), echocardiogram (ultrasound test showing the pumping action of the heart, thickness of the heart walls, and any valve leakage), and a detailed neurological examination, including maneuvers such as copying a drawing and putting pegs in a board. Patients' parents are asked questions about how they feel their child's disease affects the child's quality of life.
* Magnetic resonance imaging (MRI) to examine the heart muscle and blood flow to the heart. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The patient lies on a table that is moved into the doughnut-shaped MRI scanner, wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. A catheter (plastic tube) is placed in a vein in the child's arm so that a chemical called gadolinium can be injected during the MRI study. Gadolinium brightens areas of the heart, improving the ability to see the heart and blood flow.
* Physical medicine and rehabilitation evaluations to test the child's physical functioning. These tests include gait evaluation, measurements of the ability to exert and maintain a constant force, assessment of visual-motor control and fine motor control, aerobic exercise endurance testing, and measurement of the ability of the child's heart and lungs to increase their effectiveness with exercise.
* Idebenone/placebo treatment. Patients are given a 6-month supply of either idebenone pills or placebo (pills that look like the study drug but have no active ingredient) to take three times a day. Patients are seen by their primary care physician after 1 and 3 months on the study medication for a brief physical examination. In addition, they have blood and urine tests once a month while on medication to check for any abnormalities.
* 6-month examination. After 6 months on the study drug, patients return to NIH to repeat all the tests listed above to determine the effects of idebenone treatment.

DETAILED DESCRIPTION:
Background: Friedreich's ataxia (FA) is a progressive, autosomal recessive, multisystem degenerative disease for which there is currently no effective treatment. Recent studies have suggested that lipid-soluble antioxidants lead to a modest reversal of cardiomyopathy in patients with FA. It is possible that antioxidants may also prevent the progression of neurodegeneration.

Objective: This will be a 6 month phase 2 double-blind, placebo-controlled trial to assess the safety and efficacy of idebenone administered to adolescents and children with FA.

Study Population: We aim to enroll 48 subjects composed of children (ages 9-11) and adolescents (ages 12-17) with FA divided evenly among 4 treatment arms (placebo, low, intermediate, and high dose idebenone).

Design: Our primary objective is to examine the change in the level of oxidative stress by measuring the oxidative marker 8-hydroxy-2-deoxyguanosine from baseline and after 6 months of treatment with placebo or varying doses of idebenone. Following informed consent and assent, patients will undergo an initial medical history and physical followed by specific neurological, functional, and cardiac testing over a two-day outpatient visit. Patients will provide blood and urine samples for safety laboratory and biochemical analysis. Each patient will be randomized to one of 4 treatment arms and will be provided with a 6 month supply of study drug or placebo which will be administered three times a day. Patients will have follow-up laboratory monitoring after 1 and 3 months and at the end of the study. Additionally, patients will also have an EKG, vital signs, including orthostatics, and a physical examination performed after 1 and 3 months by their primary care physician. Patients will return after 6 months for follow-up exam, testing, and laboratory monitoring over a two-day outpatient visit.

Outcome Parameters: The primary endpoint in this phase 2 trial is the change in the level of the oxidative stress marker 8-hydroxy-2-deoxyguanosine. Secondary endpoints include types and frequency of adverse events, if any, compliance with the dosing regimen, and measurements of the following: International Cooperative Ataxia Rating Scale (ICARS), Friedreich's ataxia Rating Scale (FARS), force control, gait analysis, quantitative sensation testing, fine motor control, health related quality of life score (SF-10), functional capacity, aerobic capacity, left ventricular wall mass, noninvasive measures of systolic and diastolic ventricular function, metabolic markers, markers of mitochondrial DNA damage, and gene expression profiling.

Future Directions: We hope that the results of this phase 2 study will assist us in developing a multi-center, double-blinded, placebo-controlled phase III trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of FA with confirmed FRDA mutations.

Age from nine up to but not over eighteen years.

Weight between 30 to 80 kilograms.

Ambulatory (assistance devices permitted).

Willing to participate in all aspects of trial design and follow-up.

All subjects agree and commit to the use of 2 reliable methods of birth control for the duration of the study if sexually active.

Neurologically symptomatic.

No exposure to idebenone, coenzyme Q10, or other dietary supplements for a period of at least one month before enrollment in the study.

EXCLUSION CRITERIA:

History of a hypersensitivity reaction to idebenone or coenzyme Q10.

Pregnant or lactating women. All women of child-bearing potential must have negative serum pregnancy prior to the medication phase of the study. If a minor has a positive pregnancy test, we will inform her but not inform her parents unless we are asked to by the minor.

Platelet count, white blood cell count or hemoglobin below the lower limit of normal.

Alkaline phosphatase, SGOT, or SGPT greater than 1.5 times the upper limit of normal. Bilirubin greater than 1.5 g/dl.

Creatinine greater than 1.5 times the upper limit of normal based upon the pediatric reference range provided by the testing laboratory.

Clinically significant medical disease that, in the judgment of the investigators, would expose the patient to undue risk of harm or prevent the patient from completing the study.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2005-09-27; Primary Completion 2007-12-17 (Actual); Study Completion 2007-12-17 (Actual)

PRIMARY OUTCOMES:
To examine the change in the level of oxidative stress by measuring the oxidative marker 8-hydroxy-2-deoxyguanosine from baseline and after 6 months of treatment with placebo or varying doses of idebenone | baseline and after 6 months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of idebenone | baseline and after 6 months
To explore the effects of idebenone on cardiac parameters | baseline and after 6 months
To explore the effects of idebenone on neurological function | baseline and after 6 months
To assess the effects of idebenone on patients quality of life | baseline and after 6 months
To explore the effects of idebenone on functional capacity | baseline and after 6 months
To evaluate metabolic alterations, gene expression changes and markers of mitochondrial DNA damage | baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Fischbeck, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Harding AE. Friedreich's ataxia: a clinical and genetic study of 90 families with an analysis of early diagnostic criteria and intrafamilial clustering of clinical features. Brain. 1981 Sep;104(3):589-620. doi: 10.1093/brain/104.3.589. PMID 7272714
- [Background] Durr A, Cossee M, Agid Y, Campuzano V, Mignard C, Penet C, Mandel JL, Brice A, Koenig M. Clinical and genetic abnormalities in patients with Friedreich's ataxia. N Engl J Med. 1996 Oct 17;335(16):1169-75. doi: 10.1056/NEJM199610173351601. PMID 8815938
- [Background] Hewer RL. Study of fatal cases of Friedreich's ataxia. Br Med J. 1968 Sep 14;3(5619):649-52. doi: 10.1136/bmj.3.5619.649. PMID 5673214
- [Derived] Drinkard BE, Keyser RE, Paul SM, Arena R, Plehn JF, Yanovski JA, Di Prospero NA. Exercise capacity and idebenone intervention in children and adolescents with Friedreich ataxia. Arch Phys Med Rehabil. 2010 Jul;91(7):1044-50. doi: 10.1016/j.apmr.2010.04.007. PMID 20599042
- [Derived] Haugen AC, Di Prospero NA, Parker JS, Fannin RD, Chou J, Meyer JN, Halweg C, Collins JB, Durr A, Fischbeck K, Van Houten B. Altered gene expression and DNA damage in peripheral blood cells from Friedreich's ataxia patients: cellular model of pathology. PLoS Genet. 2010 Jan 15;6(1):e1000812. doi: 10.1371/journal.pgen.1000812. PMID 20090835
- [Derived] Di Prospero NA, Baker A, Jeffries N, Fischbeck KH. Neurological effects of high-dose idebenone in patients with Friedreich's ataxia: a randomised, placebo-controlled trial. Lancet Neurol. 2007 Oct;6(10):878-86. doi: 10.1016/S1474-4422(07)70220-X. PMID 17826341